CLINICAL TRIAL: NCT07075523
Title: Comprehensive Neuroimaging and Molecular Biomarkers of Neurotoxicity Following CAR T-Cell Therapy
Brief Title: Neuroimaging and Biomarkers of Neurotoxicity After Chimeric Antigen Receptor T-Cell Therapy
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kathryn Tringale, Assistant Professor, University of California, San Diego
Other Study IDs: 811868
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: CAR T-Cell Therapy
Keywords: CAR T-cell therapy; RBANS; ICANS; Magnetic resonance imaging
MeSH Terms: interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chimeric antigen receptor T-cell therapy: Patients recommended to undergo commercial CAR T-cell therapy
  Interventions: Other: Brain magnetic resonance imaging, neurocognitive assessments, quality of life questionnaire, biomarkers

INTERVENTIONS:
Other: Brain magnetic resonance imaging, neurocognitive assessments, quality of life questionnaire, biomarkers — Pathognomonic magnetic resonance imaging; neurocognitive assessments with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS); quality of life assessment with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30; measurement of liquid biomarkers.

SUMMARY:
The goal of this study is to understand why some people receiving chimeric antigen receptor (CAR) T-cell therapy for cancer experience neurotoxicity. The main question it aims to answer is:

Can a novel tool be developed to identify early the patients who will develop immune effector cell-associated neurotoxicity syndrome (ICANS, also called neurotoxicity) after chimeric antigen receptor (CAR) T-cell therapy?

Participants already scheduled for chimeric antigen receptor (CAR) T-cell therapy as part of the medical care for their cancer will be evaluated with advanced neuroimaging techniques. In addition, neurocognitive assessments using questionnaires and measurement of biomarkers in blood (liquid biomarkers) will be performed to provide a comprehensive characterization of neurotoxicity following chimeric antigen receptor T-cell therapy.

Assessments will be performed in the acute phase (2 to 14 days after chimeric antigen receptor (CAR) T-cell therapy) and after approximately 3 months.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm study that aims to develop a novel tool for early identification of immune effector cell-associated neurotoxicity syndrome (ICANS) in patients undergoing chimeric antigen receptor (CAR) T-cell therapy for cancer.

ICANS, which is often referred to as neurotoxicity, is a syndrome affecting the brain and the nervous system. It can give headache, confusion, difficulty concentrating, lack of energy, agitation, tremors, difficulty with language, and seizures. Up to 70% of patients undergoing chimeric antigen receptor T-cell therapy experience this neurotoxicity syndrome. Although it typically resolves within the first month after chimeric antigen receptor T-cell therapy, some patients may develop delayed or long-lasting neurological problems.

In this study, the investigators will perform a comprehensive evaluation of participants undergoing chimeric antigen receptor T-cell therapy to study neurotoxicity. The study will use advanced neuroimaging techniques of brain magnetic resonance imaging; neurocognitive assessments; evaluation of quality of life; and blood collection to measure blood-based biomarkers. Biomarkers may be measured also in cerebrospinal fluid, if collected.

To obtain a comprehensive evaluation of brain activity, 3 different brain magnetic resonance imaging modalities will be employed: T1-post-contrast, T2/FLAIR, and diffusion-weighted sequences. In addition, resting state functional magnetic resonance imaging will be performed at the baseline visit and 3 months after chimeric antigen receptor T-cell therapy.

The magnetic resonance imaging data will be applied to 3D, U-Net-based convolutional neural network that is well-validated for the detection and segmentation of brain white matter hyperintensities. The convolutional neural network magnetic resonance imaging segmentation will be integrated with neurocognition and biomarkers data to develop a model for the diagnosis of ICANS that is more quantitative and standardized compared to the current qualitative standard.

The features of neurotoxicity identified by the convolutional neural network will be correlated with biomarkers and neurocognition to evaluate the association between these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Age ≥ 18 years
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Patients recommended to undergo commercial chimeric antigen receptor T-cell therapy

Exclusion Criteria:

* Contraindication for magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see eligibility criteria
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Principal component analysis (PCA) | 2 weeks
  To identify relevant variables within three main domains (tumor imaging, neurocognitive assessments, and liquid biomarkers) collected acutely after chimeric antigen receptor (CAR) T-cell therapy that reflect distinct signatures associated with the presence of immune effector cell-associated neurotoxicity syndrome (ICANS).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Tringale, MD, MAS, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No